CLINICAL TRIAL: NCT04370652
Title: Medical Treatment of Peyronie's Disease With Collagenase Clostridium Histolyticum (CCH or Xiapex®): Sexual and Psychological Impact and Results From 156 Patients' Questionnaires Data
Brief Title: Medical Treatment of Peyronie's Disease With Collagenase Clostridium Histolyticum
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0202
Record Dates: First submitted 2020-04-15; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Peyronie Disease
Keywords: Collagenase Clostridium Histolyticum; Xiapex®; Peyronie's Disease Questionnaire (PDQ); Sexual dysfunction
MeSH Terms: conditions — Penile Induration; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peyronie's disease is the appearance of a fibrosis plaque on the albuginea of the corpora cavernosa, which produces mechanical traction at the time of erection, inducing a deformation/curvature of the erect penis. The physiopathology is largely unknown.

There is a significant sexual and psychological impact on patients. Historically, the only possible treatment was surgical. The only drug treatment that was FDA approved for this disease was Collagenase from Clostridium Histolyticum marketed under the name Xiapex® until 31/12/2019 by Sobi laboratory. Marketing was stopped on that date for economic reasons and restricted to the US market only.

The investigators propose a retrospective evaluation of the largest French monocentric series of this treatment from the perspective of the sexual and psychological evaluation of patients.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years old
* Peyronie's disease stable for more than 3 months after 12 to 18 months of evolution
* Angle of penis deformation ≥ 30°

Exclusion criteria:

* Surgery for Peyronie's disease before
* Anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peyronie's disease stable for more than 3 months after 12 to 18 months of evolution
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Peyronie's Disease Questionnaire (PDQ) | every 4 weeks for 2 years
  Peyronie's Disease Questionnaire (PDQ) : Change in baseline Peyronie's Disease Questionnaire Score each 4 weeks, i.e. before each new injection ; for up 2 years

SECONDARY OUTCOMES:
Penile curvature angulation | every 4 weeks for 2 years
  Penile curvature angulation : Change in baseline penile curvature angulation each 4 weeks, i.e. before each new injection ; for up 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Fortier, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC